CLINICAL TRIAL: NCT06025344
Title: A Single Dose Oral Bioavailability Study of PanCytoVir™ Oral Suspension (100 mg/ml) 1000 mg Versus Probenecid 500 mg Tablets, 1000 mg (2 X 500 mg) in Healthy, Adult, Human Subjects Under Fasting Conditions
Brief Title: A Relative Bioavailability Study With a Novel PanCytoVir™ Oral Suspension (100 mg/ml)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TrippBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VRS-23-002
Record Dates: First submitted 2023-08-24; First posted 2023-09-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Relative Bioavailability
MeSH Terms: interventions — Suspensions; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PanCytoVir™ 1000 mg (100 mg/mL) (Experimental): PanCytoVir™ oral suspension (100 mg/mL)
  Interventions: Drug: PanCytoVir™ 100 mg/mL oral suspension
- Probenecid 1000 mg (2x500 mg tablets) (Experimental): Probenecid 500 mg tablets
  Interventions: Drug: Probenecid 500 mg

INTERVENTIONS:
Drug: PanCytoVir™ 100 mg/mL oral suspension — Single oral dose of 1000 mg (100 mg/mL) under fasted conditions
  Arms: PanCytoVir™ 1000 mg (100 mg/mL)
Drug: Probenecid 500 mg — Single oral dose of 1000 mg under fasted conditions
  Arms: Probenecid 1000 mg (2x500 mg tablets)

SUMMARY:
An open-label, balanced, randomized, two-treatment, two-sequence, two-period, crossover, single dose oral relative bioavailability study of a novel PanCytoVir™ oral suspension (100 mg/mL) versus probenecid 500 mg tablets in normal healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy adult human subjects.
2. Subjects who are willing to participate and give informed consent
3. Subjects who are ≥ 18 years of age to ≤ 45 years of age and have a Body Mass Index between ≥18.5 to ≤ 30.0 kg/m2 extremes included, with weight of at least 50 kg.
4. Subjects with normal findings as determined by baseline history, physical examination and vital sign examination (blood pressure, pulse rate, respiration rate and body temperature).
5. Subjects with clinically acceptable findings as determined by haemogram, biochemistry, urine analysis, 12 lead ECG and chest X-ray.
6. Willingness to follow the protocol requirements especially abstaining from xanthine containing food or beverages (chocolates, tea, coffee or cola drinks) or grapefruit juice, any alcoholic products, the use of cigarettes and the use of tobacco products for 72.00 hours prior to dosing until after the last blood sample collection in each study period and adherence to food, fluid and posture restrictions.
7. No history of significant alcoholism.
8. Subject who have estimated glomerular filtration rate (eGFR) value is >60ml/min.
9. Found negative in Alcohol test.
10. Found negative in urine test for drug abuse [Benzodiazepines, Barbiturates, Morphine, Cocaine, Amphetamines and Tetrahydrocannabinol (THC)].
11. Non-smokers, ex-smokers and moderate smokers will be included. "Moderate smokers are defined as someone smoking 10 cigarettes or less per day, ex-smokers are someone who completely stopped smoking for at least 3 months."

Exclusion Criteria:

1. History of allergic responses or hypersensitivity to Probenecid or other related drugs, or any of its ingredients.
2. Requiring medication for any ailment having enzyme-modifying activity in the previous 21 days, prior to dosing day.
3. Subjects who have taken prescription medications or over-the-counter products (including vitamins and minerals) within 14 days prior to administration of study drug.
4. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
5. History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, haematological, gastrointestinal, endocrine, immunological or psychiatric diseases.
6. Participation in a clinical drug study or bioequivalence study 90 days prior to period I dosing of the present study.
7. History of malignancy or other serious diseases.
8. Blood donation 90 days prior to period I dosing of the present study.
9. Subjects with positive HIV tests, HBsAg or Hepatitis-C tests.
10. History of problem in swallowing tablets/capsules/ Suspension.
11. Any contraindication to blood sampling.
12. Female subjects found positive serum (β) Beta- hCG (Human Chorionic Gonadotropin) test.
13. Lactating women (currently breast feeding).
14. Female subjects not confirming to using birth control measures, from the date of screening until the completion of the study. Abstinence, barrier methods (condom, diaphragm, etc.) are acceptable.
15. Use of hormonal contraceptives either oral or implants.
16. History of urinary retention, gastric retention and other severe decreased gastrointestinal motility conditions, uncontrolled narrow-angle glaucoma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Bioavailability comparison using Cmax | 7 days
Bioavailability comparison using AUC | 7 days

SECONDARY OUTCOMES:
The incidence rates of AEs, TEAEs and Serious Adverse Events (SAEs) | 7 days
  Numbers and incidence rates of AEs, TEAEs and Serious Adverse Events (SAEs) will be tabulated using available version of Medical Dictionary for Regulatory Activities (MedDRA) preferred term (PT), system organ class (SOC), severity and relationship. A patient having the same AE will be counted only once in calculating frequency while patient having same AE with different start date then both will be considered for calculating frequency. If AE is with same start date but different criteria (severity, relationship to study medication and outcome), worst case/latest case (whichever applicable) will be considered. Incidence of AEs will be summarized with count (%).

CONTACTS AND LOCATIONS:
Overall Officials: David E Martin, PharmD, Study Director — TrippBio, Inc.
Locations (1):
- Vayam Research Solutions Limited, Gujrāt, India

IPD SHARING:
Plan to Share IPD: No
Plans are currently under development